CLINICAL TRIAL: NCT06784570
Title: Impact of Perioperative Levosimendan on Patients Undergoing Cardiac Surgery With Low Ejection Fraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohamed Ibrahim Mohamed El Anwar, assis professor, Zagazig University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZU-IRB # 737/15-oct-2024
Record Dates: First submitted 2025-01-12; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Surgery; Low Ejection Fraction
Keywords: levosemindan- low ejection fraction-cardiac surgery
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Intervention Model Description: patients divided into three groups according to type of surgery done : CABG alone, Valve alone and combined each group contains 80 patients, then each previous group is subdivided into LEVO group and TRAD group each subgroup contain 40 patients according to the type of inotropes used in each group either levosemindane (pre operative ) or other traditional adrenergic drugs :adrenaline ,noradrenaline ,dopamine and dobutamine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- levosemindan (Experimental): this group of patients will recieve levosemindan
  Interventions: Drug: levosemindan
- traditional (Active Comparator): this group of patients will recieve traditional intropic drugs
  Interventions: Drug: adrenaline,noreadrenaline,dopamine and doputamine

INTERVENTIONS:
Drug: levosemindan — In common practice the loading dose is omitted as it is associated with hypotension.9 Usual dose range: 0.05 to 0.2 microg/kg/min. Dose based on actual body weight up to a maximum of 120 kg.5 Commence infusion at 0.05 microg/kg/min. If the initial rate is tolerated, consider increasing the maintenance rate to 0.1 microg/kg/min after 60 minutes. If the patient remains haemodynamically stable, further increase the dose to 0.2 microg/kg/min for the remainder of the infusion.
  Arms: levosemindan
Drug: adrenaline,noreadrenaline,dopamine and doputamine — adrenaline:*4 9 %$ 0 ****8*4* 9 : ,- 4 - *4 9 * C % F*4 9 9 9 noreadrenaline:# *4 9 C % 9 F 9 9 *4* Q*4 9 9 dopamine:9 * C % 9 F 9 9 ) * 9 9 dobutamine:9 * C % F 9 9 9 * 9 9
  Arms: traditional

SUMMARY:
to compar levosemindan to other cardiac intropic medications that strengthen the heart in diffrent common adult heart surgery with patients with low ejection fraction(weak heart)

DETAILED DESCRIPTION:
in this study show the effect of levosemindan use during coronary artery surgery ,heart valve surgery and combined coronary and valve surgery in comparison to other traditional medications with patients with low ejection fraction(weak heart)

ELIGIBILITY:
Inclusion Criteria:

1. Valve surgery
2. CABG surgery,
3. combined surgery
4. all patients Ejection Fraction less than 35 ٪ -

Exclusion Criteria:

1. Patients age ≤ 20-70 < years
2. Aortic and redo surgery
3. any patients with Ejection Fraction more than 35 ٪ -

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
death through day 30, | 1 month (no scale for measurement as death may occured due to multible causes that be difficult to be identified and measured )
  death occured either intraoperative , ICU, ward or after discharge to home within month of the day of the surgery
Renal-replacement therapy | 1 month
  included haemodialysis, peritoneal dialysis, or continuous Veno venous haemodialysis(indicated when serum creatinine above 2.0 mg/dl or an increase of 50% above baseline value)
Perioperative myocardial infarction | 5 days
  defined as a creatine kinase MB level of more than 100 ng per millilitre or a level that was more than 10 times the upper limit of the normal range specified at the local laboratory, regardless of changes on the electrocardiogram, or a creatine kinase MB level that was more than 50 ng per millilitre or a level that was more than 5 times the upper limit of the normal range with new Q waves that were more than 30 msec in duration in two contiguous leads or new left bundle-branch block
Intra Aortic Ballon Pumb insertion | 5 days(no scale for measurement )
  it consisidered to be one of the ventricular assissted device that need to be inserted in post cardiac surgery shocked patiients that not respond heamdynamically to highest doses of cardiac intropes

CONTACTS AND LOCATIONS:
Locations (1):
- cardiothorathic surgery department -faculty of medecine-zagazig univeristy-Egypt, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No